CLINICAL TRIAL: NCT03815266
Title: Feasibility Study to Evaluate the Observance Rehabilitation of Upper Limbs by Visual-motor Simulation Associated at Transcranial Direct Current Stimulation (tDCS) in Hemiparetic Patient Post-stroke.
Acronym: SIMSTIM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped due to lack of inclusions
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1708098; 2018-A01883-52 (Other: ANSM)
Record Dates: First submitted 2018-11-06; First posted 2019-01-24 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Stroke
Keywords: transcranial Direct Current Stimulation (tDCS); Computerized Mirror Therapy (CMT); hemiparetic; Ischemic; stroke; Intensive Visual Simulation3 (IVS3)
MeSH Terms: conditions — Stroke; Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with first ischemic or hemorrhagic stroke (Experimental): Patient with first ischemic or hemorrhagic stroke will be included. They will have the following program Computerized Mirror Therapy (CMT) associated at transcranial Direct Current Stimulation (tDCS). This program will consist of 5 sessions per week for 4 weeks (20 minutes).
  In more, they will have the following tests: Tolerance Assessment Questionnaire, Ashworth's scale, Frenchay arm test, Abilhand questionnaire, Fugl-Meyer test, and Goal Attainment Scaling (GAS).
  Interventions: Diagnostic Test: transcranial Direct Current Stimulation (tDCS); Diagnostic Test: Computerized Mirror Therapy (CMT); Diagnostic Test: Tolerance Assessment Questionnaire; Diagnostic Test: Ashworth's scale; Diagnostic Test: Frenchay arm test; Diagnostic Test: Abilhand questionnaire; Diagnostic Test: Fugl-Meyer test; Diagnostic Test: Goal Attainment Scaling (GAS)

INTERVENTIONS:
Diagnostic Test: transcranial Direct Current Stimulation (tDCS) — transcranial Direct Current Stimulation (tDCS) is device which consist in setting up an electrode on the skull of the patient to deliver the low intensity current.
  Patient will have transcranial Direct Current Stimulation (tDCS) at each session and at the same time of Computerized Mirror Therapy (CMT).
Diagnostic Test: Computerized Mirror Therapy (CMT) — Computerized Mirror Therapy (CMT) will be realizing by the device Intensive Visual Simulation 3 (IVS3). Patient will have Computerized Mirror Therapy (CMT) at each session and at the same time of transcranial Direct Current Stimulation (tDCS).
  Other Names: Intensive Visual Simulation3 (IVS3)
Diagnostic Test: Tolerance Assessment Questionnaire — The Tolerance Assessment Questionnaire will be completed at the end of each session.
Diagnostic Test: Ashworth's scale — Ashworth's scale evaluates the resistance to stretching. This test will be completed before the start of the program, at the end of the program and one month after.
Diagnostic Test: Frenchay arm test — Frenchay arm test evaluates your abilities with the affected hand to perform several actions.
  This test will be completed before the start of the program, at the end of the program and one month after.
Diagnostic Test: Abilhand questionnaire — Abilhand questionnaire evaluates your abilities to perform several activities in the daily life with your arm affected.
  This test will be completed before the start of the program, at the end of the program and one month after.
Diagnostic Test: Fugl-Meyer test — Fugl-Meyer test evaluates your ability to perform different movements with all the joints of your arm affected.
  This test will be completed before the start of the program, at the end of the program and one month after.
Diagnostic Test: Goal Attainment Scaling (GAS) — Goal Attainment Scaling (GAS) sets therapeutic goals with the patient before the start of the program.
  These goals will be checked at the end of the program and one month after.

SUMMARY:
Although the mirror therapy is recognized as effective, its practice is difficult, especially with hemiplegic patients. It is difficult for them to understand, control the movements and carry out a double task with the two upper limbs. The implementation of a Computerized Mirror Therapy (CMT) with the Intensive Visual Simulation 3 (IVS3) device makes it possible to limit these problems by proposing pre-recorded sessions, not limited to the right or left hemi-space, and proposing a work on proximal motricity. Since the functional prognosis of the upper hemiplegic limb remains mostly unfavourable, a wide range of interventions should be proposed. There is currently a consensus to consider the use of transcranial Direct Current Stimulation (tDCS) stimulation in functional recovery after stroke as a method to enhance the effectiveness of training techniques. Although all motor therapies can theoretically benefit from increased effectiveness by the addition of transcranial Direct Current Stimulation (tDCS), Computerized Mirror Therapy (CMT) has a high potential for sensitivity to transcranial Direct Current Stimulation (tDCS) due to the intensity of the motor training of the upper limb applied.

DETAILED DESCRIPTION:
The primary objective of this study is to investigate the feasibility of a program combining Computerized Mirror Therapy (CMT) with dual- transcranial Direct Current Stimulation (tDCS) stimulation by evaluating observance to hemiparetic stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient with first ischemic or hemorrhagic stroke for less than one year, having not recidivated since then and responsible for initially complete left or right hemiplegia
* Modified Frenchay arm test score <70 (/ 100)
* Without a neurological history other than stroke
* Having signed the written consent and affiliated or entitled to a social security scheme

Exclusion Criteria:

* Patient with contraindications to transcranial Direct Current Stimulation (tDCS) or Transcranial Magnetic Stimulation (TMS) (brain metal implant, pacemaker, other implanted active medical device)
* Patient who didn't have cerebral Magnetic Resonance Imaging (MRI) imaging during their stroke
* With complete lesion of the primary motor cortex
* With alcohol / drug dependence
* With psychiatric illness, cognitive impairment, uncontrolled disease / epilepsy, malignant disease, severe renal or pulmonary disease
* With a history of disabling associated disease
* With cerebellar syndrome
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2022-04-14 (Actual)

PRIMARY OUTCOMES:
Rate of observance of the program Computerized Mirror Therapy (CMT) + transcranial Direct Current Stimulation (tDCS) | Up to Day 40
  Rate of observance of the program CMT + tDCS. It is will be measured by the number of patients who will be finished the study.

SECONDARY OUTCOMES:
Effect of the program Computerized Mirror Therapy (CMT) + transcranial Direct Current Stimulation (tDCS) improving activities of the upper limb - measured by Frenchay arm test | Day 40
  To evaluate the effect of the program Computerized Mirror Therapy (CMT) + transcranial Direct Current Stimulation (tDCS) improving activities of the upper limb.
  It is will be measured by Frenchay arm test.
Effect of the program Computerized Mirror Therapy (CMT) + transcranial Direct Current Stimulation (tDCS) improving activities of the upper limb - measured by Frenchay arm test | Day 70
  To evaluate the effect of the program Computerized Mirror Therapy (CMT) + transcranial Direct Current Stimulation (tDCS) improving activities of the upper limb.
  It is will be measured by Frenchay arm test.
occurrence of epileptic seizure | Day 40
  Measure of tolerance of the program Intensive Visual Simulation 3 (IVS3) + transcranial Direct Current Stimulation (tDCS) by the occurrence of epileptic seizure report by adverse event and serious adverse events.
occurrence of Anxiety crisis | Day 40
  Measure of tolerance of the program Intensive Visual Simulation 3 (IVS3) + transcranial Direct Current Stimulation (tDCS) by the occurrence of anxiety crisis report by adverse event and serious adverse events.
Tolerance Assessment Questionnaire | Up to day 70
  Analysis the results of the Tolerance Assessment Questionnaire.
Evaluation of the program by Goal Attainment Scaling (GAS) | Day 40
  Analysis of evaluation of the program by Goal Attainment Scaling (GAS) results.
Evaluation of the program by Goal Attainment Scaling (GAS) | Day 70
  Analysis of evaluation of the program by Goal Attainment Scaling (GAS) results.
Quantitative improvement of the deficiencies - Fugl-Meyer test | Day 40
  Measure of the quantitative improvement of the deficiencies by analysis of Fugl-Meyer test results.
Quantitative improvement of the deficiencies - Fugl-Meyer test | Day 70
  Measure of the quantitative improvement of the deficiencies by analysis of Fugl-Meyer test results.
Abilities to perform several activities - Abilhand questionnaire | Day 40
  Analysis of abilities to perform several activities in the daily life by Abilhand questionnaire results.
Abilities to perform several activities - Abilhand questionnaire | Day 70
  Analysis of abilities to perform several activities in the daily life by Abilhand questionnaire results.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal GIRAUX, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No